CLINICAL TRIAL: NCT00572091
Title: An Open-Label, Single-Arm Pilot Study of the Safety and Efficacy of the Percutaneous Transvenous Mitral Annuloplasty Device Used to Reduce Mitral Regurgitation
Brief Title: Aachen Safety and Efficacy of the Percutaneous Transvenous Mitral Annuloplasty Device to Reduce Mitral Regurgitation
Acronym: PTOLEMY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Viacor (Industry)
Responsible Party: Katharine M Stohlman, Viacor, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-055P
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Heart Failure; Mitral Regurgitation
Keywords: Heart Failure; Mitral Regurgitation
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patient is screened for study and given baseline assessments. Patient receives a diagnostic PTMA assessment and if responsive, receives a PTMA implant.
  Interventions: Device: PTMA Implant

INTERVENTIONS:
Device: PTMA Implant — Percutaneous assessment from right or left subclavian vein, with PTMA implant in the coronary sinus, great cardiac vein.

SUMMARY:
Improvement in heart failure with moderate to severe mitral regurgitation using a percutaneously delivered implanted device

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure
* functional MR 2+ - 4+
* LVEF 20% - 50%

Exclusion Criteria:

* MR of organic origins
* significant co-morbidities

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-02; Primary Completion 2008-04 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
percent of patients who remain free from device-related major adverse events: death, myocardial infarction, tamponade, emergent cardiac surgery | 30 days

SECONDARY OUTCOMES:
percent of implanted patients who maintain a sustained 1 grade reduction in mitral regurgitation and reduction in mitral anterior posterior dimension | 30 days
improvement of clinical symptoms of heart failure as defined by percent of implanted patients who exhibit one of the following: decrease in NYHA class, improvement in Minnesota QOL survey, increase in 6 minute walk, improvement in VO2 max. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Hoffmann, MD, Principal Investigator — Rheinisch-Westfalische Technische Hochschule, Universitätsklinikum Aachen
Locations (1):
- Rheinisch-Westfalische Technische Hochschule, Universitätsklinikum Aachen, Aachen, Germany